CLINICAL TRIAL: NCT04963309
Title: Extubation in the Operating Room After Living Donor Liver Transplantation in Adult Patients: a Retrospective Observational Study
Brief Title: Extubation in the Operating Room After Living Donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Clinical associate professor, Pusan National University Yangsan Hospital
Other Study IDs: 05-2021-052
Record Dates: First submitted 2021-06-29; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Extubation in the OR After LDLT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OR-EX: the group with endotracheal tube extubation in the operating room in patients who underwent living-donor liver transplantation for end-stage liver failure
  Interventions: Other: endotracheal tube extubation in the operating room
- NOR-EX: the group without endotracheal tube extubation in the operating room in patients who underwent living-donor liver transplantation for end-stage liver failure

INTERVENTIONS:
Other: endotracheal tube extubation in the operating room — endotracheal tube extubation in the operating room
  Groups: OR-EX

SUMMARY:
Duration of mechanical ventilation, length of intensive care unit stay, length of postoperative hospital stay, and the incidence rates of complications between the group with endotracheal tube extubation in the operating room (OR-EX) and those without (NOR-EX) in patients who underwent living-donor liver transplantation for end-stage liver failure are going to be compared. Through these results, it is investigated whether endotracheal tube extubation in the operating room is useful in reducing the length of stay in the intensive care unit and the hospital stay after surgery in patients who have undergone living-donor liver transplantation.

DETAILED DESCRIPTION:
Long-term mechanical ventilation after liver transplantation may increase the risk of complications such as pneumonia, sepsis, and multi-organ failure. Recent advances in surgical techniques and the introduction of short-acting anesthetics have accelerated the recovery of liver transplant recipients, and early extubation after liver transplantation is being proposed as a standard method. The results of a study on early extubation in patients undergoing liver transplantation suggested a reduction in the length of stay in the neutralizer room and predictors of early extubation. However, these studies are limited to males, and there is no study in which the definition of early extubation includes extubation in the operating room or extubation in the operating room within 1-3 hours of arrival in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older who underwent living-donor liver transplantation for end-stage liver failure

Exclusion Criteria:

* A score of 26 or higher on the model for end-stage liver disease (MELD) scale
* In case of endotracheal intubation when entering the operating room
* If hepatic encephalopathy is stage 3 or higher at the time of admission to the operating room
* When the arterial blood partial pressure (PaO2)/inhaled oxygen fraction (FiO2) ratio is less than 200 on the Arterial Blood Gas Analysis (ABGA) before the end of the living liver transplantation operation
* Preoperative chest X-ray examination or chest computed tomography shows pulmonary edema
* If patients is diagnosed with hepatopulmonary syndrome before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients 18 years of age or older who underwent living-donor liver transplantation for end-stage liver failure
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
length of intensive care unit stay | during intensive care unit stay, up to 3 months
  length of intensive care unit stay
length of postoperative hospital stay | during hospital stay, up to 6 months
  length of postoperative hospital stay

SECONDARY OUTCOMES:
incidence rates of complications | during admission, up to 6 months
  incidence rates of complications

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea